CLINICAL TRIAL: NCT00137839
Title: A Phase II Study of Erlotinib (OSI-774); Tarceva in Women With Previously Untreated Advance Adenocarcinoma of the Lung
Brief Title: Erlotinib in Women With Previously Untreated Adenocarcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pasi A. Janne, MD, PhD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pasi A. Janne, MD, PhD, Associate Professor, Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-253
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Adenocarcinoma; Non-small Cell Lung Cancer
Keywords: Tarceva; Erlotinib; OSI-774; Adenocarcinoma; Advanced Lung Cancer
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erlotinib (Experimental): Erlotinib: 150 mg orally once daily without interruption Cycle duration considered 4 weeks and treatment duration indefinite until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Tarceva; OSI-774

SUMMARY:
The purpose of this trial is to figure out what effects (good or bad) the investigational drug agent called Tarceva (erlotinib; OSI-774) has on women with previously untreated adenocarcinoma.

DETAILED DESCRIPTION:
Patients will start taking Tarceva daily by mouth on Day 1 and will continue taking this medication daily at home, until participation in the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of adenocarcinoma of the lung
* Patient has had at least one core biopsy of her tumor
* Must be willing to undergo epidermal growth factor receptor (EGFR) mutation testing of her tumor
* Stage four (IV) or three (III) B non-small cell lung cancer
* Non-smoker or former smoker. Non-smoker is defined as a person who smoked 100 or less cigarettes in her lifetime while a former smoker is defined as a person who has quit smoking one or more years ago.
* Three or more weeks since last radiation therapy
* Three or more weeks since last major surgery
* Must at least be able to walk and capable of taking care of herself although unable to carry out work activities
* Life expectancy of 8 weeks or more
* Blood tests that show kidneys, liver and bone marrow to be working adequately
* Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the entire time enrolled in study

Exclusion Criteria:

* Prior exposure to Tarceva (OSI-774, erlotinib)
* Uncontrolled central nervous system problems
* Prior chemotherapy regimen
* Difficulty swallowing
* A disease or disorder that interferes with ability to digest and absorb food
* Incomplete healing of previous oncologic or other major surgery
* Significant medical history or unstable medical condition such as heart failure, active infection, uncontrolled high blood pressure
* Pregnant or breast feeding
* A medical condition that could make it unsafe for patient to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Perez-Soler R, Chachoua A, Hammond LA, Rowinsky EK, Huberman M, Karp D, Rigas J, Clark GM, Santabarbara P, Bonomi P. Determinants of tumor response and survival with erlotinib in patients with non--small-cell lung cancer. J Clin Oncol. 2004 Aug 15;22(16):3238-47. doi: 10.1200/JCO.2004.11.057. PMID 15310767
- [Background] Janne PA, Engelman JA, Johnson BE. Epidermal growth factor receptor mutations in non-small-cell lung cancer: implications for treatment and tumor biology. J Clin Oncol. 2005 May 10;23(14):3227-34. doi: 10.1200/JCO.2005.09.985. PMID 15886310
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- See also: Dana-Farber Cancer Institute Lowe Thoracic Oncology Program — https://www.dana-farber.org/thoracic-lung-cancer-treatment-center/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled November 2004 to November 2008.
Period: Overall Study
Arm/Group | Erlotinib
Started | 84
Treated | 83
Completed | 0 (Data on Reason Not Completed reflects Reason Off-Study)
Not Completed | 84
Not completed — Adverse Event | 7
Not completed — Physician Decision | 7
Not completed — Death | 8
Not completed — Disease Progression | 60
Not completed — Not Start Treatment | 1
Not completed — Prolonged Treatment Delay | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 84
Age, Continuous [Mean (Full Range); unit: years] — Population: One participant was missing date of birth information.
  years
    number analyzed (Participants) | 83
    (all) | 65 [34 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 78
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 84
EGFR Status [Count of Participants; unit: Participants] — Mutation status in the epidermal growth factor receptor (EGFR) gene in tumor specimens was determined by standard methods of immunohistochemistry.
  Participants
    Wild Type | 36
    Mutant | 39
    Unevaluable | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieve partial response (PR) or better on treatment based on RECIST 1.0 criteria: For target lesions, complete response (CR) is disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD (both require a minimum of 4 weeks). Progressive disease (PD) is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or appearance of one or more new target lesions. Stable disease (SD) is neither PR nor PD. For non-target lesions, PD is the appearance of one or more new non-target lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: In this study cohort, treatment duration which parallels the maximum observation time was up to 39 months.
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 83
percentage of participants | 27.7 [18.5 to 38.7]

2. Secondary Outcome: Overall Response Rate (ORR) by EGFR Mutation Status
Description: ORR is defined as the percentage of participants who achieve partial response (PR) or better on treatment based on RECIST 1.0 criteria: For target lesions, complete response (CR) is disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD (both require a minimum of 4 weeks). Progressive disease (PD) is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or appearance of one or more new target lesions. SD is neither PR nor PD. For non-target lesions, PD is the appearance of one or more new non-target lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: In this study cohort, treatment duration which parallels the maximum observation time was up to 39 months.
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- EGFR Mutant: Mutation status of the epidermal growth factor receptor (EGFR) gene in tumor specimens was determined by standard methods of immunohistochemistry.
- EGFR Wild Type; Unevaluable EGFR: Mutation status in the epidermal growth factor receptor (EGFR) gene in tumor specimens was determined by standard methods of immunohistochemistry.
Arm/Group | EGFR Mutant | EGFR Wild Type | Unevaluable EGFR
Number analyzed (Participants) | 39 | 35 | 9
percentage of participants | 56.4 [39.6 to 72.2] | 2.9 [0.1 to 12.8] | 0.0 [0.0 to 33.6]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from study entry to death or date last known alive.
Time Frame: In this study cohort, participants were followed for survival up to 155 months.
Population: The analysis dataset is comprised of all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 84
months | 22.9 [15.7 to 26.5]

4. Secondary Outcome: Overall Survival by EGFR Mutation Status
Description: OS is defined as the time from study entry to death or date last known alive.
Time Frame: In this study cohort, participants were followed for survival up to 155 months.
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGFR Mutant | EGFR Wild Type | Unevaluable EGFR
Number analyzed (Participants) | 39 | 36 | 9
months | 32.6 [24.4 to 44.0] | 9.9 [6.6 to 16.2] | 15.7 [1.4 to 109.6]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) based on the National Cancer Institute's Common Toxicity Criteria for Adverse Events version 3 (CTCAEv3) were assessed every 4 weeks on treatment. In this study cohort, treatment duration which parallels the maximum observation time was up to 39 months.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.The analysis dataset for AEs is comprised of all treated participants versus all enrolled for all cause mortality/any death on study.
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 83/84
Serious Adverse Events (participants affected / at risk) | 33/83
Other Adverse Events (participants affected / at risk) | 83/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=83)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 5
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 5
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 4
Extremity-lower (gait/walking) (General disorders) | 4
Liver dysfunction/failure (Hepatobiliary disorders) | 4
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 4
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 4
Infection Gr0-2 neut, skin (Infections and infestations) | 4
INR (Investigations) | 3
PTT (Investigations) | 3
ALT, SGPT (Investigations) | 4
AST, SGOT (Investigations) | 4
Bilirubin (Investigations) | 4
Creatinine (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 4
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 14
Skin-other (Skin and subcutaneous tissue disorders) | 5
Thrombosis/thrombus/embolism (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=83)
Death - disease progression NOS (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 12
Hematologic-other (Blood and lymphatic system disorders) | 5
DIC (Blood and lymphatic system disorders) | 4
Palpitations (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 5
Sinus tachycardia (Cardiac disorders) | 5
Arrhythmia-other (Cardiac disorders) | 5
C-P arrest, non-fatal, cause unknown (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 5
Valvular heart disease (Cardiac disorders) | 5
Cardiac-other (Cardiac disorders) | 7
External ear, pain (Ear and labyrinth disorders) | 4
Hyopthyroidism (Endocrine disorders) | 5
Dry eye syndrome (Eye disorders) | 15
Ocular surface disease (Eye disorders) | 3
Vision-blurred (Eye disorders) | 4
Tearing (Eye disorders) | 3
Ocular-other (Eye disorders) | 4
Eye, pain (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 11
Dentures or dental prosthesis (Gastrointestinal disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 62
Dry mouth (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 10
Hemorrhoids (Gastrointestinal disorders) | 5
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 13
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 26
Proctitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 13
GI-other (Gastrointestinal disorders) | 5
Anus, hemorrhage (Gastrointestinal disorders) | 5
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 5
Rectum, hemorrhage (Gastrointestinal disorders) | 5
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 5
Pancreatitis (Gastrointestinal disorders) | 5
Abdomen, pain (Gastrointestinal disorders) | 6
Oral cavity, pain (Gastrointestinal disorders) | 4
Oral gums, pain (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 33
Fever w/o neutropenia (General disorders) | 5
Rigors/chills (General disorders) | 3
Constitutional, other (General disorders) | 5
Death - multiorgan failure (General disorders) | 1
Death - sudden death (General disorders) | 1
Edema limb (General disorders) | 6
Extremity-lower (gait/walking) (General disorders) | 4
Chest/thoracic pain NOS (General disorders) | 12
Pain NOS (General disorders) | 4
Pain-other (General disorders) | 6
Liver dysfunction/failure (Hepatobiliary disorders) | 4
Allergic reaction (Immune system disorders) | 5
Infection w/ gr3-4 neut, wound (Infections and infestations) | 4
Infection Gr0-2 neut, external ear (Infections and infestations) | 4
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 4
Infection Gr0-2 neut, lip/perioral (Infections and infestations) | 4
Infection Gr0-2 neut, lung (Infections and infestations) | 4
Infection Gr0-2 neut, nerve-periph (Infections and infestations) | 4
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 4
Infection Gr0-2 neut, skin (Infections and infestations) | 6
Infection Gr0-2 neut, stomach (Infections and infestations) | 4
Infection Gr0-2 neut, ungual (Infections and infestations) | 4
Infection Gr0-2 neut, upper airway (Infections and infestations) | 7
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 4
Infection Gr0-2 neut, vagina (Infections and infestations) | 4
Infection Gr0-2 neut, wound (Infections and infestations) | 4
Infection w/ unk ANC conjunctiva (Infections and infestations) | 4
Infection w/ unk ANC dental-tooth (Infections and infestations) | 4
Infection w/ unk ANC lymphatic (Infections and infestations) | 4
Infection w/ unk ANC middle ear (Infections and infestations) | 4
Infection w/ unk ANC nose (Infections and infestations) | 4
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 4
Infection w/ unk ANC pharynx (Infections and infestations) | 4
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 4
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 4
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 4
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 5
Infection w/ unk ANC vagina (Infections and infestations) | 4
Infection w/ unk ANC wound (Infections and infestations) | 4
Infection Gr 0-2 neut, blood (Infections and infestations) | 4
Infection-other (Infections and infestations) | 6
Bruising (Injury, poisoning and procedural complications) | 2
Burn (Injury, poisoning and procedural complications) | 5
Fracture (Injury, poisoning and procedural complications) | 5
Leukocytes (Investigations) | 5
Neutrophils (Investigations) | 5
Platelets (Investigations) | 5
Weight loss (Investigations) | 9
INR (Investigations) | 3
PTT (Investigations) | 3
Coagulation-other (Investigations) | 5
Alkaline phosphatase (Investigations) | 8
ALT, SGPT (Investigations) | 11
AST, SGOT (Investigations) | 12
Bilirubin (Investigations) | 19
Creatinine (Investigations) | 5
Metabolic/Laboratory-other (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 23
Dehydration (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 5
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 5
Back, pain (Musculoskeletal and connective tissue disorders) | 6
Bone, pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 4
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 9
Joint, pain (Musculoskeletal and connective tissue disorders) | 7
Muscle, pain (Musculoskeletal and connective tissue disorders) | 5
Neck, pain (Musculoskeletal and connective tissue disorders) | 4
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Taste disturbance (Nervous system disorders) | 16
Cognitive disturbance (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 11
Encephalopathy (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 5
Neuropathy CN VII face-motor / taste (Nervous system disorders) | 5
Neuropathy-sensory (Nervous system disorders) | 7
Depressed level of consciousness (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 4
Neurologic-other (Nervous system disorders) | 5
Ocular-other (Nervous system disorders) | 11
Head/headache (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 9
Confusion (Psychiatric disorders) | 5
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 6
Proteinuria (Renal and urinary disorders) | 5
Obstruction-urethra (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 3
Renal/GU-other (Renal and urinary disorders) | 5
Breast, pain (Reproductive system and breast disorders) | 4
Vaginal dryness (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 5
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 5
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 8
Apnea (Respiratory, thoracic and mediastinal disorders) | 3
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 4
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 7
Sweating (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 47
Alopecia (Skin and subcutaneous tissue disorders) | 21
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 17
Photosensitivity (Skin and subcutaneous tissue disorders) | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 23
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 66
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 5
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 4
Ulceration (Skin and subcutaneous tissue disorders) | 4
Skin-other (Skin and subcutaneous tissue disorders) | 36
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 5
Hot flashes (Vascular disorders) | 3
Hematoma (Vascular disorders) | 5
Hemorrhage-other (Vascular disorders) | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No